CLINICAL TRIAL: NCT01588899
Title: China Clinical Trial for Therapeutic MRI-guided High Intensity Focused Ultrasound Ablation of Uterine Fibroids
Brief Title: China Clinical Trial for Therapeutic MR-HIFU Ablation of Uterine Fibroids
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philips Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 907764
Record Dates: First submitted 2012-04-27; First posted 2012-05-01 (Estimated); Last update posted 2015-10-22 (Estimated); Status verified 2015-10

CONDITIONS: Uterine Fibroids
Keywords: Uterine Leiomyomas; Fibroids; HIFU; Ablation; High Intensity Focused Ultrasound
MeSH Terms: conditions — Leiomyoma; Myofibroma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MR-HIFU Treatment (Experimental): Patients in this arm will receive MR-HIFU uterine fibroid treatment
  Interventions: Device: MR-HIFU uterine fibroid treatment

INTERVENTIONS:
Device: MR-HIFU uterine fibroid treatment — A single treatment session for uterine fibroids with the MR-HIFU device.
  Other Names: Philips Sonalleve MR-HIFU

SUMMARY:
The purpose of this study is to demonstrate safety and effectiveness of the Philips Sonalleve Magnetic Resonance Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) for treatment of uterine fibroids in a Chinese population.

DETAILED DESCRIPTION:
This study is to confirm the safety and effectiveness of Magnetic Resonance Imaging-guided High Intensity Focused Ultrasound (MR-HIFU) in ablating uterine tissue associated with symptomatic leiomyomas. The importance of this therapy is that it offers a non-invasive, uterine sparing procedure for the treatment of uterine fibroids in pre- and peri- menopausal women.

MR-HIFU uses ultrasound to heat and thermally ablate fibroid tissue. The MRI system identifies the ultrasound path and monitors heat rise in the fibroid tissue. The goal of the study is to show treatment safety and effectiveness of the Philips Sonalleve MR-HIFU device for uterine fibroids marketing approval in the Chinese market. MR-HIFU will be performed in 100 patients who pass inclusion/exclusion criteria. Safety, quality of life, and imaging endpoints will be evaluated in all study patients at baseline and at 6 months post-treatment. All patients will be followed up for 12 months post-treatment for safety.

ELIGIBILITY:
Inclusion Criteria:

* Women, age between 18 and 55 years
* Weight < 140 kg
* Pre- or peri-menopausal
* Uterine size < 24 weeks
* Cervical cell assessment by Pap smear/Thin-prep Cytologic Test (TCT): Normal, Low Grade Squamous Intraepithelial Lesion (SIL), Low risk Human Papillomavirus (HPV) or Atypical Squamous Cells of Uncertain Significance (ASCUS) subtypes of cervical tissue
* Fibroids selected for treatment meeting the following criteria:

  1. Total planned ablation volume of all fibroids should not exceed 250 ml, and
  2. No more than 5 fibroids should be planned for ablation, and
  3. Dominant fibroid (diameter) is greater than or equal to 3 cm, and
  4. Fibroids which are completely non-enhancing under Magnetic Resonance (MR) contrast agent should not be treated as the identification of treated volume becomes ambiguous
  5. Highly perfused or brighter than myometrium in T2-weighted MRI (according to the T2 contrast obtained using the Philips MR-HIFU protocol) fibroids should not be treated
* MR-HIFU device accessibility to fibroids such that at least 50% of the total fibroid volume can be treated
* Willing and able to attend all study visits

Exclusion Criteria:

* Other pelvic disease (Other mass, endometriosis, ovarian tumor, acute pelvic disease, significant adenomyosis)
* Desire for future pregnancy
* Significant systemic disease, even if controlled
* Positive pregnancy test
* Hematocrit < 25%
* Extensive scarring along anterior lower abdominal wall (> 50% of area)
* Surgical clips in the direct path of the HIFU beam
* MRI contraindicated
* MRI contrast agent contraindicated
* Fibroids not quantifiable on MRI (e.g. multi-fibroid cases where volume measurements are not feasible)
* Calcifications around or throughout uterine tissues
* Communication barrier
* Suspected malignancy

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 107 (Actual)
Dates: Start 2012-05; Primary Completion 2014-12 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change in fibroid volume | At baseline and at 6 months after treatment
  Proportion of patients with treated fibroid volume at 6 months after treatment reduced to 90% or less of treated fibroid volume at baseline (before MR-HIFU treatment)
Adverse Events | Within 6 months after treatment
  Number of Adverse Events reported as resulting from MR-HIFU treatment

CONTACTS AND LOCATIONS:
Overall Officials: Qinping Liao, Principal Investigator — Peking University First Hospital; Yueling Wang, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (2):
- China (2):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - First Affiliated Hospital of Medical College of Xi'an Jiaotong University, Xi'an

REFERENCES:
- [Derived] Chen R, Keserci B, Bi H, Han X, Wang X, Bai W, Wang Y, Yang X, Yang J, Wei J, Seppala M, Viitala A, Liao Q. The safety and effectiveness of volumetric magnetic resonance-guided high-intensity focused ultrasound treatment of symptomatic uterine fibroids: early clinical experience in China. J Ther Ultrasound. 2016 Nov 3;4:27. doi: 10.1186/s40349-016-0072-9. eCollection 2016. PMID 27822376